CLINICAL TRIAL: NCT03945370
Title: Oral Ketone Body Supplementation in Patients With McArdle Disease
Acronym: GSDV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, Principle investigator, MD, research fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18033230.1
Record Dates: First submitted 2019-02-18; First posted 2019-05-10 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: McArdle Disease
MeSH Terms: conditions — Glycogen Storage Disease Type V

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, single-blind, cross-over study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention sequence 1 (Active Comparator): Ketone drink first - Placebo drink secondly
  Interventions: Dietary Supplement: β-hydroxybuturate esters; Dietary Supplement: Placebo drink
- Intervention sequence 2 (Placebo Comparator): Placebo drink first - Ketone drink secondly
  Interventions: Dietary Supplement: β-hydroxybuturate esters; Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: β-hydroxybuturate esters — Oral dietary supplement product containing β-hydroxybuturate esters
Dietary Supplement: Placebo drink — Oral placebo drink

SUMMARY:
McArdle disease, glycogen storage disease type V, is a rare metabolic disease. Affected individuals are unable to utilize sugar stored as glycogen in muscle.

Investigators hypothesize that ketones can be an alternative fuel substrate for skeletal muscle when muscle glycogenolysis is blocked as in McArdle disease.

In this study investigators will investigate the immediate effects of an oral supplementation of exogenous ketone bodies (poly-hydroxybuturate) on exercise capacity in patients with metabolic myopathies, compared with a placebo drink.

DETAILED DESCRIPTION:
McArdle disease, glycogen storage disease type V, is a rare metabolic disease caused by mutations in the PYGM gene resulting in absence of the enzyme muscle phosphorylase. Affected individuals are unable to utilize sugar stored as glycogen in muscle, leading to exercise intolerance, exercise-induced muscle pain, contractures and rhabdomyolysis, which may cause renal failure. Currently, there are no satisfactory treatment options for McArdle disease.

A key element of alleviating symptoms in McArdle disease is to provide alternative fuels for energy metabolism. Investigators hypothesize that ketones can be an alternative fuel substrate for skeletal muscle when muscle glycogenolysis is blocked as in McArdle disease.

Aim: To investigate the immediate effects of an oral supplementation of exogenous ketone bodies (poly-hydroxybuturate) on exercise capacity in patients with metabolic myopathies.

Supplement description: food supplement containing β-hydroxybuturate esters

Methods:

Study design: Placebo-controlled, single-blind, cross-over study. Inclusion: 5-8 patients with McArdle disease and 3-5 healthy controls.

Time table:

Subjects will meet to 2 test days. Subjects will be randomized using a 1:1 assignment ratio to receive either the keto-drink or placebo drink first. The oral supplement received will be blinded for the participants and the investigators. On each test day, subjects spend approximately 4 hours at the laboratory:

* Insertion of peripheral brachial venous catheters for extracting blood samples and stable isotope infusion and hydroxybutyrate infusion.
* Baseline blood sampling, medical examination, vital sign measurements, weight and height.
* Stable isotope infusion 2 hours before the cycling exercise test. Three stable isotope tracers [2,4-13C2]-D- β-hydroxybutyrate, [1,1,2,3,3-2H5]-glycerol and [6,6-2H2]-glucose solutions, are infused via a venous catheter until a steady-state is reached. The tracer infusions will continue during the cycling test. The tracers (all from Cambridge Isotope Laboratories, Andover, MA, USA) will be dissolved and injected into a solution of 0.9% saline (NaCl) through a bacterial filter.
* One Ketone or placebo drink administration 30 minutes before the exercise test
* Subjects will perform a 40 minutes cycle exercise test at a constant load corresponding to 60-70% of their VO2max (found in a screening study). During the test, subjects wear a mask for continuous gas-exchange measurements and ECG electrodes to determine VO2 and heart rate during constant load cycling (VO2const and HRconst). Blood samples will be drawn 4 times before, every 10 minutes during exercise and after exercise. During the test participants will be asked to rate perceived exertion (RPE) on a Borg scale.

ELIGIBILITY:
Inclusion criteria:

* Genetically confirmed McArdle disease or healthy control.
* Patient is willing and able to provide written informed consent prior to participation.
* Patient is ambulatory.

Exclusion criteria:

* Patient has any prior or current medical conditions that, in the judgment of the Investigator, would prevent the patient from safely participating in and/or completing all study requirements.
* Pregnancy or breastfeeding
* Patient does not have the cognitive capacity to understand/comprehend and complete all study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Heart rate | 30 minuts x 2
  Change between visit 1 and 2 in mean heart rate during constant load cycling exercise (40 minute submaximal cycle test)

SECONDARY OUTCOMES:
Ketone metabolism | 150 minuts x 2
  Change between visit 1 and 2, measured with stable isotope technique during the constant load cycling test
Carbohydrate metabolism | 150 minuts x 2
  Change between visit 1 and 2, measured with stable isotope technique during the constant load cycling test
Fat metabolism | 150 minuts x 2
  Change between visit 1 and 2, measured with stable isotope technique during the constant load cycling test
Indirect calorimetry | 30 minuts x 2
  Changes in oxidation rates at visit 1 and visit 2, measured via indirect calorimetry before and during exercise
Perceived exertion | 30 minuts x 2
  Changes in perceived exertion beween visit 1 and 2 during the cycle test
Blood ketone | 150 minuts x 2
  Changes in ketone bodies in the blood between visit 1 and 2, measured at both before, during and at end exercise.
Insulin | 30 minuts x 2
  Insulin changes between visit 1 and 2 measured before, during and at end exercise.
Metabolites | 30 minuts x 2
  changes between visit 1 and 2

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No